CLINICAL TRIAL: NCT03753191
Title: The Effects of Transcranial Direct Current Stimulation on Executive Function in People With Mild to Moderate Dementia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Frank LAI, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: StartUp1.51
Record Dates: First submitted 2018-11-17; First posted 2018-11-26 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Dementia; Executive Function; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Dementia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: double-blinded, randomized case-control interventional study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blinded, with randomized case-control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- People with Dementia (Experimental): Twenty subjects each group will be randomized to receive either anodal tDCS or shame tDCS over the Right iFG or Left DLPFC. A 2mA direct current for active tDCS (current density : .057 mA/cm2) with a 20 mins stimulation period
  Interventions: Device: transcranial direct current stimulation
- Health Control (Sham Comparator): Twenty subjects each group will be randomized to receive either anodal tDCS or shame tDCS over the Right iFG or Left DLPFC. After a fade in period of 10s to mimic initial tDCS peripheral skin sensations, the stimulator will be turned off in order to prevent the induction of any neuromodulatory effect.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — Each subject will undergo one tDCS stimulation session lasting for 20 minutes. A constant current of 2 mA will be applied with a linear fade in, fade out of 10 seconds to prevent electrical transients.

SUMMARY:
To study the effects of transcranial direct current stimulation on executive function in people with mild to moderate dementia

DETAILED DESCRIPTION:
Extensive research had shown executive dysfunction in people with dementia (PWD) is associated with functional abnormalities in prefrontal regions such as the right inferior frontal gyrus (Right IFG) or the left dorsal lateral pre-frontal cortex (Left DLPFC) . Clinical studies suggest that tDCS may be a useful therapeutic tool. Post-tDCS improvements have also been shown in visuo-motor coordination of healthy controls and performance in working memory. The aim of this study is to investigate the effect of tDCS stimulation over left DLPFC or right IFG on attention, inhibition and working memory and their neural correlates in people with dementia (PWD) and healthy controls (HC).This study is planned as a double-blinded, randomized case-control interventional study with a duration of 30 months.

ELIGIBILITY:
Inclusion Criteria:

* PWD must be aged at least 65 years or above when informed consent is obtained in the presence of his / her first degree relatives.
* PWD must meet criteria of DSM-V for dementia as well as for historical diagnosis of dementia.
* PWD must have a Chinese MoCA score > 19 (mild to moderate cognitive deficits) at screening.
* Subjects (both PWD and HC) must be physically healthy, and must be able to understand and be willing to sign the informed consent document

Exclusion Criteria:

* Subject with major neurological illness.
* Subject with other diagnosed psychiatric disorders
* Subjects reported with history of substance abuse, which including alcohol, drugs or any medication which is indicative of chronic abuse.
* Failures to comply with the study protocol or to follow the instructions.
* Self-reported with known skin diseases or skin allergy history.
* Self-reported with metallic implants, dentures
* Self-reported with history of claustrophobia. (This is excluded because subject needs to stay in a quiet room with the head-mounted fNIRS and tDCS, which may elicit their feeling of anxiety)

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-10-20 (Estimated)

PRIMARY OUTCOMES:
Haemodynamic changes | baseline and 5 minutes after tDCS
  Change in hemodynamic level in two region of interest of prefrontal cortical regions, that is DLPFC and IFG
Trail Making Test | baseline and 5 minutes after tDCS
  change in Trail Making Test
Behavior change | baseline and 5 minutes after tDCS
  Change in the Chinese Multiple Errands Test
N-back task | baseline and 5 minutes after tDCS
  Change in N-back task
Stop-signal task | baseline and 5 minutes after tDCS
  Change in Stop-signal task

CONTACTS AND LOCATIONS:
Overall Officials: Frank LAI, PhD, Principal Investigator — Assistant Professor
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nitsche MA, Paulus W. Sustained excitability elevations induced by transcranial DC motor cortex stimulation in humans. Neurology. 2001 Nov 27;57(10):1899-901. doi: 10.1212/wnl.57.10.1899. PMID 11723286
- [Background] Liebetanz D, Nitsche MA, Tergau F, Paulus W. Pharmacological approach to the mechanisms of transcranial DC-stimulation-induced after-effects of human motor cortex excitability. Brain. 2002 Oct;125(Pt 10):2238-47. doi: 10.1093/brain/awf238. PMID 12244081
- [Result] Antal A, Varga ET, Kincses TZ, Nitsche MA, Paulus W. Oscillatory brain activity and transcranial direct current stimulation in humans. Neuroreport. 2004 Jun 7;15(8):1307-10. doi: 10.1097/01.wnr.0000127460.08361.84. PMID 15167555
- [Result] Zaehle T, Sandmann P, Thorne JD, Jancke L, Herrmann CS. Transcranial direct current stimulation of the prefrontal cortex modulates working memory performance: combined behavioural and electrophysiological evidence. BMC Neurosci. 2011 Jan 6;12:2. doi: 10.1186/1471-2202-12-2. PMID 21211016